CLINICAL TRIAL: NCT05811598
Title: Random、Control and Open Study of Real Word Study on Myopia Control With Repeated Red Light Therapy for Ages of 3~6 Years Old
Brief Title: Real Word Study on Myopia Control With Repeated Red Light Therapy for Ages of 3~6 Years Old
Acronym: RMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Airdoc Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beijing Airdoc Technology Co.,
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Myopia; Amblyopia
Keywords: Myopia; Children; LLLT; PBM
MeSH Terms: conditions — Myopia; Amblyopia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: two groups for the 2 lighting lever (0.37mW and 0.6mW）for 2 groups of ages (3~4 years old and 5~6 years old)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repeated red light therapy for 3~4 year-old myopia (Experimental): 0.37mW lighting with wavelength of 650nm for the age of 3~4 years old(including both 3 and 4 years)myopia.
  Interventions: Device: repeated ultra low lever red light
- repeated red light therapy for 5~6 year-old myopia (Experimental): 0.60mW lighting with wavelength of 650nm for the age of 5~6 years old(including both 5 and 6 years)myopia.
  Interventions: Device: repeated ultra low lever red light

INTERVENTIONS:
Device: repeated ultra low lever red light — Myopia indoor lighting therapy
  Other Names: LLLT, PBM therapy

SUMMARY:
Repeated Red Light Therapy had been used as an amblyopia therapy for children as well as the myopia control in primary schools. However, ultra low lever of red light therapy with irradiance of 0.37mW and 0.60mW effectiveness and safety for 3~ 6 year-old myopia treatment or slow myopia progression are seldom reported.

DETAILED DESCRIPTION:
Repeated Red Light Therapy had been used as an amblyopia therapy for children as well as the myopia control in primary schools. However, ultra low lever of red light therapy with irradiance of 0.37mW and 0.60mW effectiveness and safety for 3~ 6 year-old myopia treatment or slow myopia progression are seldom reported. Here we design this control and random prospective study to find the two types light with different irridance to two ages (3~4 years old and 5~6 years old) respectively. Wether the dose and effectiveness exit or not for 3~6- year- old myopia control.

ELIGIBILITY:
Inclusion Criteria:

* 3~6 years old;
* Myopia Spherical Equivalence Refraction <=-0.50D;
* Written Informed Consent;

Exclusion Criteria:

* Cannot approval with written informed consent;
* Photophobia or allergy to red light;
* With other severe conditions the principle investigators refused to enroll this study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean changes of axial length vaules by millimeter at follow-up from baseline. | at 3-month and at 6-month
  Ocular axial length measured by IOLmaster500 or Lenstar will be measured and recorded at follow-ups and at baseline. The changes values of axial length of both groups will be compared as the main outcome to compare the effectiveness of repeated red light thearpy.

SECONDARY OUTCOMES:
Numbers of children without myopic refraction changes by spherical equivalence values from refraction at follow-up from baseline(D) | at 3-month and at 6-month
  Cycloplegic refraction changes from baseline will be measured and recorded at follow-up and at baseline. Spherical equivalence will be calculated with the formular of SE=spherical diopter+1/2cylinder diopter
Number of Participants with unsafety issues during the study | at 6-month
  Adverse event and device failure rate

OTHER OUTCOMES:
Rate of subjects meet with repeated red light thearpy greater than 85% of the specified requirementsfrequence record | at 1-month, 3-month and 6-month
  Twice daily with an interval of 4 hours or mor, and 3 minutes at each session

CONTACTS AND LOCATIONS:
Overall Officials: Chao He, PhD, Study Director — Beijing Airdoc Technology Co., Ltd.; Daoman Xiang, MD, PhD, Principal Investigator — Guangzhou Women and Children's Medical Center; Wensi Shen, MD, PhD, Study Chair — Guangzhou Women and Children's Medical Center
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided